CLINICAL TRIAL: NCT01224483
Title: Multicenter Retrospective Analysis About the Clinical Characteristics of Korean Patients With PNH
Brief Title: Multicenter Retrospective Analysis About the Clinical Characteristics of Korean Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Jun Ho Jang, Aplastic Working Party, The Korean Society of Hematology
Other Study IDs: 2010-02-048
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Hemoglobinuria, Paroxysmal
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Paroxysmal nocturnal hemoglobinuria (PNH) is a hematopoietic stem cell disorder in which unregulated activation of the complement system leads to significant ischemic morbidities with shortened lifespan. Life-threatening thromboembolism (TE) is the most feared complication of PNH, accounting for up to 45% of patient deaths. It is estimated that 40% of PNH patients experience a clinically evident TE and 60% of patients without clinically diagnosed TE demonstrate TE by high-sensitivity MRI, indicating the ongoing thrombotic risk in most patients with PNH. Much of these data come from PNH patients from European descent. To understand the impact of TE in patients with PNH from non-European regions, we performed this study to evaluate the clinical characteristics of Korean patients with PNH.

DETAILED DESCRIPTION:
To evaluate the clinical characteristics in Korean PNH patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis confirmed by Ham's test or Flow cytometry Patients have any Flow cytometry data

Exclusion Criteria:

* Patients have no Flow cytometry data

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean PNH patients: diagnosis confirmed by Ham's test or Flow cytometry
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Jang, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Division of Hematology Oncology, Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jang JH, Kim JS, Yoon SS, Lee JH, Kim YK, Jo DY, Chung J, Sohn SK, Lee JW. Predictive Factors of Mortality in Population of Patients with Paroxysmal Nocturnal Hemoglobinuria (PNH): Results from a Korean PNH Registry. J Korean Med Sci. 2016 Feb;31(2):214-21. doi: 10.3346/jkms.2016.31.2.214. Epub 2016 Jan 26. PMID 26839475
- [Derived] Kim JS, Jang JH, Yoon SS, Lee JH, Kim YK, Jo DY, Chung JS, Sohn SK, Lee JW. Distinct subgroups of paroxysmal nocturnal hemoglobinuria (PNH) with cytopenia: results from South Korean National PNH Registry. Ann Hematol. 2016 Jan;95(1):125-133. doi: 10.1007/s00277-015-2511-z. Epub 2015 Sep 29. PMID 26416513
- [Derived] Lee JW, Jang JH, Kim JS, Yoon SS, Lee JH, Kim YK, Jo DY, Chung J, Sohn SK. Clinical signs and symptoms associated with increased risk for thrombosis in patients with paroxysmal nocturnal hemoglobinuria from a Korean Registry. Int J Hematol. 2013 Jun;97(6):749-57. doi: 10.1007/s12185-013-1346-4. Epub 2013 May 1. PMID 23636668